CLINICAL TRIAL: NCT04089488
Title: Prospective Observational Study of Site-Specific Incident and Prevalent Cases of Cancer in People Living With HIV/AIDS- in Latin America
Brief Title: Incidence and Prevalence of Cancer in People Living With HIV/AIDS at Cancer Centers in Latin America
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-S008; NCI-2019-01734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-S008 (Other: AIDS Malignancy Consortium); AMC-S008 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: HIV Infection; Human Immunodeficiency Virus 1 Positive; Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — HIV Infections; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (respond to surveys, medical record review): Patients respond to surveys and/or undergo medical record review at baseline and at 4 weeks.
  Interventions: Other: Medical Chart Review; Other: Survey Administration

INTERVENTIONS:
Other: Medical Chart Review — Correlative studies
  Other Names: Chart Review
Other: Survey Administration — Respond to surveys

SUMMARY:
This trial studies the frequency of incident and prevalent of cancer in people living with human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS) at cancer centers in Latin America. By counting how many people living with HIV/AIDS have cancer at these specific centers, researchers may better understand how they are being treated and cared for. This may help researchers to understand what new studies may be helpful for those areas in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the number of diagnosed cancers in people living with HIV/AIDS (PLWHA) presenting to participating clinical sites in Latin America, and estimate site-specific prevalence based on all presenting cancers (new diagnosis, recurrence, and surveillance cases) and site-specific incidence based on newly diagnosed cancers.

SECONDARY OBJECTIVES:

I. Obtain information on the use of diagnostic testing and treatment for the cohort of diagnosed HIV-associated cancer participants.

II. To collect information on participant characteristics for diagnosed HIV-associated cancers (e.g., antiretroviral therapy [ART] regimen, current CD4 count, current viral load, etc.).

OUTLINE:

Patients respond to surveys and/or undergo medical record review at baseline and at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive. Documentation of HIV-1 infection by means of any one of the following:

  * Documentation of receipt of ART by a licensed health care provider (Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name);
  * HIV-1 ribonucleic acid (RNA) detection by a licensed HIV-1 RNA assay demonstrating > 1000 RNA copies/mL, and confirmed by a licensed screening antibody and/or HIV antibody/antigen combination assay;
  * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay, such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay.
  * Note: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally.
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/Custom Industrial Analysis (CIA) that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* Must have a current or prior (within the last 5 years) diagnosis of cancer, but there is no restriction of the number or type of prior treatments. Participants will qualify under one of three categories:

  * New diagnosis: no prior treatment for current malignancy. May be prior to, or currently receiving the first line of therapy.
  * Prior diagnosis (within 5 years), in remission: Not currently on cancer treatment other than combination antiretroviral therapy (cART). Prior treatment for malignancy can include surgery, radiation, or chemotherapy (or cART initiation in Kaposi sarcoma [KS]). No restriction on number of prior lines of therapy.
  * Prior diagnosis, recurrent: considering or currently receiving treatment that is not first line. No restriction on the number of prior lines of therapy.
* Date of birth and age should be determined based on best possible information or documentation available.
* Ability to understand and the willingness to provide informed consent document.

Exclusion Criteria:

* Participants not meeting all criteria above are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants presenting to HIV treatment programs or cancer treatment programs at collaborating sites, with both HIV and cancer, which may include either a history of malignancy or current diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Strother, Principal Investigator — AIDS Malignancy Consortium
Locations (4):
- Hospital de Agudos Juan A. Fernandez, Buenos Aires, Argentina
- Brazil (2):
  - Instituto Nacional de Câncer José de Alencar, Rio de Janeiro
  - Complexo Hospitalar Universitário Professor Edgard Santos, Salvador
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Started | 175
Completed | 175
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 167
  >=65 years | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [33 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 171
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 47
  More than one race | 0
  Unknown or Not Reported | 100
Region of Enrollment [Number; unit: participants]
  Argentina | 26
  Brazil | 49
  Mexico | 100

OUTCOME MEASURES:

1. Primary Outcome: Estimates of Site-specific Incident Cases and Site-specific Prevalence of Cases Presenting With Human Immunodeficiency Virus (HIV) and Cancer Presenting Over 9 Months at the Clinical Sites
Description: The primary endpoint will be the estimates of site-specific frequency of new diagnosis and existing cases (recurrence and surveillance) presenting with HIV and cancer presenting over 1 year, 9 months (21 months) at the clinical sites.
Time Frame: Up to 21 months
Population: There are five study sites (Complexo Hospitalar; Hospital Fernandez; Hospital Roff0; Instituto Nacional De Cancer Brazil ; and Instituto de Oncologia). Given a study site, new diagnosis and existing cases(recurrence and surveillance) are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Participants
  Complexo Hospitalar Professor Edgard Santos (new diagnosis) | 13
  Complexo Hospitalar Professor Edgard Santos (recurrence) | 4
  Complexo Hospitalar Professor Edgard Santos (surveillance) | 10
  Hospital Fernandez (new diagnosis) | 10
  Hospital Fernandez (recurrence) | 2
  Hospital Fernandez (surveillance) | 5
  Hospital Roffo (new diagnosis) | 3
  Hospital Roffo (recurrence) | 2
  Hospital Roffo (surveillance) | 4
  Instituto Nacional De Cancer Brazil (new diagnosis) | 11
  Instituto Nacional De Cancer Brazil (recurrence) | 2
  Instituto Nacional De Cancer Brazil (surveillance) | 9
  Instituto de Oncologia (new diagnosis) | 27
  Instituto de Oncologia (recurrence) | 9
  Instituto de Oncologia (surveillance) | 64

2. Primary Outcome: Mean Cases Per Month of New Cases Were Estimated Along With Corresponding 95% Poisson Confidence Interval by Study Site.
Description: The mean cases per month of incidence will be estimated along with corresponding 95% Poisson confidence interval. The number of cases will be counted and mean cases per months will be estimated. Duration of observation was 21 months.
  This summary was based on the study site.
Time Frame: 21 months
Population: There are five study sites (Complexo Hospitalar; Hospital Fernandez; Hospital Roff0; Instituto Nacional De Cancer Brazil ; and Instituto de Oncologia). Given a study site, new diagnosis cases are summarized using cases per month.
Measure: Mean (95% Confidence Interval); unit: New diagnosis cases per month
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
New diagnosis cases per month
  Complexo Hospitalar Professor Edgard Santos (new diasgnosis): number analyzed (Participants) | 27
  Complexo Hospitalar Professor Edgard Santos (new diasgnosis) | 0.62 [0.33 to 1.06]
  Instituto Nacional De Cancer Brazil (new diagnosis): number analyzed (Participants) | 22
  Instituto Nacional De Cancer Brazil (new diagnosis) | 0.52 [0.26 to 0.94]
  Instituto de Oncologia (new diagnosis): number analyzed (Participants) | 100
  Instituto de Oncologia (new diagnosis) | 1.29 [0.84 to 1.87]
  Hospital Fernandez (new diagnosis): number analyzed (Participants) | 17
  Hospital Fernandez (new diagnosis) | 0.48 [0.23 to 0.88]
  Hospital Roffo (new diagnosis): number analyzed (Participants) | 9
  Hospital Roffo (new diagnosis) | 0.14 [0.03 to 0.42]

3. Primary Outcome: Mean Cases Per Month of New Cases Were Estimated Along With Corresponding 95% Poisson Confidence Interval by Cancer Type.
Description: The mean cases per month of incidence will be estimated along with corresponding 95% Poisson confidence interval. The number of cases will be counted and mean cases per months will be estimated. Duration of observation was 21 months.
  This summary was based on the cancer type.
Time Frame: 21 months
Population: The numbers of participants per cancer type were displayed.
Measure: Mean (95% Confidence Interval); unit: Mean cases per month
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Mean cases per month
  Kaposi sarcoma (new diagnosis): number analyzed (Participants) | 70
  Kaposi sarcoma (new diagnosis) | 1.19 [0.77 to 1.75]
  Non-Hodgkin's Lymphoma (new diagnisis): number analyzed (Participants) | 46
  Non-Hodgkin's Lymphoma (new diagnisis) | 0.86 [0.51 to 1.35]
  Hodgkin's lymphoma (new diagnosis): number analyzed (Participants) | 13
  Hodgkin's lymphoma (new diagnosis) | 0.24 [0.08 to 0.56]
  Anal cancer (new diagnosis): number analyzed (Participants) | 3
  Anal cancer (new diagnosis) | 0 [0 to 0]
  Cervical cancer (new diagnosis): number analyzed (Participants) | 5
  Cervical cancer (new diagnosis) | 0.10 [0.01 to 0.34]
  Other (new diagnosis): number analyzed (Participants) | 38
  Other (new diagnosis) | 0.67 [0.36 to 1.12]

4. Primary Outcome: Mean Cases Per Month of Existing Cases Were Estimated Along With Corresponding 95% Poisson Confidence Interval by Study Site.
Description: The mean cases per month of prevalence will be estimated along with corresponding 95% Poisson confidence interval. The number of cases will be counted and mean cases per months will be estimated. Duration of observation was 21 months.
  This summary was based on the study site.
Time Frame: 21 months
Population: The numbers of participants per study site were displayed.
Measure: Mean (95% Confidence Interval); unit: mean cases per month
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
mean cases per month
  Complexo Hospitalar Professor Edgard Santos: number analyzed (Participants) | 27
  Complexo Hospitalar Professor Edgard Santos | .67 [.36 to 1.12]
  Instituto Nacional De Cancer Brazil: number analyzed (Participants) | 22
  Instituto Nacional De Cancer Brazil | 0.52 [0.26 to 0.94]
  Instituto de Oncologia: number analyzed (Participants) | 100
  Instituto de Oncologia | 3.48 [2.72 to 4.37]
  Hospital Fernandez: number analyzed (Participants) | 17
  Hospital Fernandez | 0.33 [0.13 to 0.69]
  Hospital Roffo: number analyzed (Participants) | 9
  Hospital Roffo | 0.29 [0.10 to 0.62]

5. Primary Outcome: Mean Cases Per Month of Existing Cases Were Estimated Along With Corresponding 95% Poisson Confidence Interval by Cancer Type
Description: The mean cases per month of prevalence will be estimated along with corresponding 95% Poisson confidence interval. The number of cases will be counted and mean cases per months will be estimated. Duration of observation was 21 months.
  This summary was based on the cancer type.
Time Frame: 21 months
Population: The numbers of participants per cancer type were displayed.
Measure: Mean (95% Confidence Interval); unit: Mean cases per month
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Mean cases per month
  Kaposi sarcoma: number analyzed (Participants) | 70
  Kaposi sarcoma | 2.14 [1.56 to 2.87]
  non-Hodgkin's Lymphoma: number analyzed (Participants) | 46
  non-Hodgkin's Lymphoma | 1.33 [0.89 to 1.93]
  Hodgkin's Lymphoma: number analyzed (Participants) | 13
  Hodgkin's Lymphoma | 0.38 [0.16 to 0.75]
  Anal cancer: number analyzed (Participants) | 3
  Anal cancer | 0.14 [0.03 to 0.42]
  Cervical cancer: number analyzed (Participants) | 5
  Cervical cancer | 0.14 [0.03 to 0.42]
  Other: number analyzed (Participants) | 38
  Other | 1.14 [0.73 to 1.70]

6. Secondary Outcome: Information on the Use of Diagnostic Testing in HIV-positive Individuals
Description: The frequency of diagnostic testing modalities will be summarized for cancer.
Time Frame: Up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Participants
  Histology (Kaposi sarcoma) | 62
  Clinical only (Kaposi sarcoma) | 7
  Histology (Non-Hodgkin's lymphoma) | 45
  Cytology (Non-Hodgkin's lymphoma) | 1
  Histology (Hodgkin's lymphoma) | 12
  Cytology (Hodgkin's lymphoma) | 1
  Histology(Anal) | 3
  Histology (Cervical) | 5
  Histology (Other) | 38
  Unknown | 1

7. Secondary Outcome: HIV Treatment and Disease Characteristics of HIV-positive Individuals Diagnosed With Cancer
Description: For each cancer, summary statistics will be used to describe the HIV treatment regimens and disease characteristics.
Time Frame: Up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Participants
  Kaposi sarcoma (NNRTI only) | 17
  Kaposi sarcoma (Combination) | 48
  Kaposi sarcoma (No HIV treatment) | 5
  Non-Hodgkin's lymphoma (NNRTI only) | 18
  Non-Hodgkin's lymphoma (Combination) | 25
  Non-Hodgkin's lymphoma (No HIV treatment) | 3
  Hodgkin's lymphoma (NNRTI only) | 4
  Hodgkin's lymphoma (Combination) | 8
  Hodgkin's lymphoma (No HIV treatment) | 1
  Anal (NNRTI only) | 1
  Anal (Combination) | 2
  Cervical (Combination) | 4
  Cervical (No HIV treatment) | 1
  Other (NNRTI only) | 21
  Other (Combination) | 12
  Other (No HIV treatment) | 5

8. Secondary Outcome: Information on the Treatment for Cancers Diagnosed in HIV-positive Individuals
Description: The frequency of the Treatment for Cancers Diagnosed in HIV-positive Individuals will be summarized.
Time Frame: Up to 21 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 175
Participants
  Surgery only | 3
  surgery and chemotherapy | 2
  Radiation only | 2
  Radiation and chemotherapy | 3
  Chemotherapy only | 24
  Chemotherapy and other | 1
  Other | 11
  No information | 129

9. Secondary Outcome: CD4 of HIV-positive Individuals Diagnosed With Cancer
Description: CD4 percent of HIV-positive Individuals Diagnosed With Cancer will be summarized.
Time Frame: Baseline
Population: 1 missing CD4 value
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 cells
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 174
Percentage of CD4 cells
  Kaposi sarcoma: number analyzed (Participants) | 69
  Kaposi sarcoma | 15 [8 to 22]
  Non-Hodgkin's lymphoma: number analyzed (Participants) | 46
  Non-Hodgkin's lymphoma | 14.5 [9 to 25]
  Hodgkin's lymphoma: number analyzed (Participants) | 13
  Hodgkin's lymphoma | 17 [16 to 24]
  Anal: number analyzed (Participants) | 3
  Anal | 18 [13 to 24]
  Cervical: number analyzed (Participants) | 5
  Cervical | 18 [16 to 24]
  Other: number analyzed (Participants) | 38
  Other | 26 [18 to 35]

10. Secondary Outcome: HIV Viral Load of HIV-positive Individuals Diagnosed With Cancer
Description: HIV viral load of HIV-positive Individuals Diagnosed With Cancer will be summarized
Time Frame: Baseline
Population: 89 participants were assessed for this Outcome Measure.
Measure: Median (Inter-Quartile Range); unit: copies per ml
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
Number analyzed (Participants) | 89
copies per ml
  Kaposi sarcoma: number analyzed (Participants) | 38
  Kaposi sarcoma | 46 [40 to 1125]
  Non-Hodgkin's lymphoma: number analyzed (Participants) | 22
  Non-Hodgkin's lymphoma | 40.5 [40 to 29246]
  Hodgkin's lymphoma49: number analyzed (Participants) | 7
  Hodgkin's lymphoma49 | 49 [40 to 364]
  Anal: number analyzed (Participants) | 2
  Anal | 30 [20 to 40]
  Cervical: number analyzed (Participants) | 2
  Cervical | 40.5 [40 to 41]
  Other: number analyzed (Participants) | 18
  Other | 40 [40 to 47]

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: No participants were assessed for deaths or adverse events.
Arm/Group | Observational (Respond to Surveys, Medical Record Review)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04089488/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT04089488/ICF_001.pdf